CLINICAL TRIAL: NCT07208188
Title: Transcutaneous Spinal Cord Stimulation for Rehabilitation of Upper Limbs in Early Spinal Cord Injury: Randomised Feasibility Study
Brief Title: tESCS for Upper Limb Rehab in Spinal Cord Injury
Acronym: SCIRUS
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); The Queen Elizabeth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN24NE012; SMSR009 (Other Grant/Funding Number: Stoke Mandeville Spinal Research)
Record Dates: First submitted 2025-09-01; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: Tetraplegia; incomplete; subacute; transcutaneous spinal cord stimulation; randmised feasibility study
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Intervention Model Description: Randomised feasibility study The study design will be a randomised double blinded feasibility study. The investigators will recruit 20 participants, equally split into active and control interventions. The active group will receive upper limb therapy with transcutaneous spinal cord stimulation (tESCS) 1 hour per day, 5 days per week, for 4 weeks, while the control group will receive the same amount of sham therapy with tESCS electrodes placed as in the active group but with only 1 minute of electrical stimulation to achieve blinding.
  Note that tESCS has a medical CE mark
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): One hour of transcutaneous electrical stimulation alongside conventional occupational therapy
  Interventions: Device: Transcutaneous spinal cord stimulation (tESCS) active group
- Control (Sham Comparator): Receiving 1 minute of stimulation alongside the conventional occupational therapy
  Interventions: Device: Sham transcutaneous spinal cord stimulation (tESCS)

INTERVENTIONS:
Device: Transcutaneous spinal cord stimulation (tESCS) active group — Participants in the active arm will receive 60 min of tESCS alongside the conventional occupation therapy, 20 sessions for 4 weeks, 5 times per week
  Arms: Intervention
Device: Sham transcutaneous spinal cord stimulation (tESCS) — The control group will receive only 1 min of tESCS while doing conventional occupational therapy for 60 min. Number of session 20, 4 weeks, 5 times a week
  Arms: Control

SUMMARY:
Regaining hand and arm function is an important step towards regaining independence following high-level spinal cord injury (tetraplegia). The delivery of small electrical pulses over the skin above the spinal cord, called transcutaneous spinal cord stimulation (tESCS), appears to improve the arm and hand function of people who have had tetraplegia for several years when delivered at the same time as upper limb therapy. However, tESCS has not been tested in people who have a new spinal cord injury. It should be straightforward to deliver tESCS during standard upper limb therapy sessions to inpatients receiving primary rehabilitation. The investigators want to test the practical aspects of delivering this intervention and also to compare recovery between a group of people who only receive upper limb therapy and a group who receive upper limb therapy and tESCS. If successful, tESCS could in the future be used as part of regular therapy following an acute spinal cord injury. Benefits could include faster and better recovery, reduced stay in hospital, and reduced NHS costs.

DETAILED DESCRIPTION:
Background Spinal Cord Injury affects more than 50,000 people in the UK, with an incidence of 2400 new cases every year. Muscular paralysis and sensory loss carry substantial physiological, psychological, financial, and social costs. Almost 60% of people affected by SCI sustain a high-level injury, that is, injury to spinal levels C2-T1, affecting arms and hands. Restoring hand and arm function is a top priority for people with tetraplegia, where even small improvements of motor function, combined with available assistive devices, may greatly improve independence and quality of life.

Transcutaneous spinal cord stimulation (tESCS) has emerged as a viable neuromodulation approach for facilitating the recovery of motor function in people with SCI. Studies that have applied tESCS at cervical segments combined with activity-based upper limb rehabilitation. Such active-assisted exercises such as gross and fine motor skill training, maximum voluntary contraction training, and unimanual and bimanual task performance have shown significant improvements in upper limb function.

It is believed that tESCS stimulation activates motor neuronal networks of the spinal cord, including the recruitment of afferent fibres in the posterior root, to elevate spinal network excitability. The underlying hypothesis is that after severe cervical SCI, nonfunctional sensory-motor networks within the cervical spinal cord can be transcutaneously neuromodulated to physiological states that enable and amplify voluntary control of the arm and hand.

A multicentre ONWARD Up-LIFT trial, which included 14 research sites, including QENSIU, has demonstrated functional improvements in people with incomplete chronic tetraplegia. As part of a UK Neuromodulation Network, we were awarded funding to deliver a substantial follow-up study, focusing on chronic complete tetraplegia. The results are showing some neurological recovery but modest functional improvement, indicating that some minimal level of preserved sensory or motor function is required in order to benefit from tESCS. For that reason, the investigators plan to recruit people with incomplete SCI in this study.

Rationale In the area of upper limb rehabilitation, the focus has been mainly on people with chronic SCI, likely due to the lack of alternative rehabilitation strategies and the difficulty in applying acute interventions in the clinical setting [3-8]. However, to date, there have been limited studies reporting the use of tESCS with people with subacute SCI. A randomised controlled trial with 22 complete or incomplete tetraplegic patients (3-12 months post injury, probably recruited from home) compared 8 sessions of tESCS with Armeo robot exercise to 8 sessions of Armeo alone. Both groups achieved comparable functional improvement but Armeo group had a higher change in scores. Our recent search of ClinTrials.gov (search criteria Spinal Cord Injuries, Upper extremity dysfunctions and electrical stimulation) has however, identified no current or future study which includes people with subacute SCI and randomisation.

There are multiple technologies for people with subacute tSCI, including robotics, functional electrical stimulation, or more recently Brain Computer interface. Then, why do the investigators need yet another rehabilitation technology? There are several features that stand tESCS apart from the other rehabilitation technologies, both when it comes to usability and the mechanism of action. Most notably tSCI facilitates performing functional movements, therefore it can be combined with the existing therapy sessions, rather than requiring extra sessions like e.g. robotic devices or having multiple precisely defined stimulation sites like FES. Setup time is much shorter and the price is lower than robotics. This is of critical importance for the clinical adoption of technology, where lack of time in busy therapists' and patients' schedules is often a major barrier to larger-scale trials that would provide solid scientific evidence.

An obvious advantage of using tESCS in the subacute rather than in the chronic stage is the potential to supplement natural recovery. In addition, unused muscle has inevitably deconditioned in chronic SCI, therefore weeks of training to optimise muscle health is preferred prior to chronic tESCS intervention, which itself necessitates a large number of sessions. In one research study, the investigators identified requirements for (accompanied) transport and travel time to and from the hospital as the main factors impeding recruitment and increasing dropout rates in chronic patients. These are not issues for patients undergoing primary rehabilitation Finally, while months of tESCS training are required to achieve improvement in people with chronic SCI, it is not known whether this time would be substantially shorter in people undergoing primary rehabilitation post SCI and whether these benefits would be long-lasting.

Answering these questions and demonstrating the feasibility of delivering tESCS integrated with standard upper limb therapy would be major steps toward adopting this technology into clinical practice.

The investigators aim to test the feasibility of delivering tESCS to hospitalised (undergoing primary rehabilitation) tetraplegic patients by combining it with standard upper limb therapy. The investigators hypothesise that tESCS will be straightforward to implement and that it will not significantly burden staff or interrupt the existing patient schedule. The investigators also hypothesise that combining tESCS with conventional upper limb therapy will result in larger functional and neurological improvements than therapy alone.

Over 60% of people sustaining spinal cord injury have tetraplegia, resulting in a high level of disability. tESCS has shown very promising results in people with chronic injuries. Based on results from these studies, the investigators believe that tESCS has the potential to result.in substantial improvement in neurological recovery if delivered in parallel with primary rehabilitation.

This study will provide the first high quality evidence of the feasibility of incorporating tESCS into clinical practice in the acute care setting. Physical therapy/activity is an essential co-therapy of tESCS By combining tESCS with standard therapy, the additional burden on therapists will be minimised, increasing the chances of successful clinical translation of the technology.

the investigators hypothesise that the positive effect of tESCS will be greater in the acute/subacute than in the chronic phase and that therefore it would be possible to see significant improvement after only a few weeks of intervention. Improved neurological function should lead to a reduced length of stay and healthcare costs. The results of this study will be the first step towards a larger multicentre trial evaluating the early use of tESCS, a vital step towards wider adoption of tESCS in clinical settings. Such clinical adoption would have the potential to benefit all people with acute tetraplegia.

The efficient delivery of tESCS and the relative affordability of the device (costing under £10K they are much cheaper than robotic devices) greatly enhance the generalisability of the results for any future clinical trial.

Theoretical Framework It is believed that tESCS stimulation activates motor neuronal networks of the spinal cord, including the recruitment of afferent fibres in the posterior root, to elevate spinal network excitability. The underlying hypothesis is that after severe cervical SCI, nonfunctional sensory-motor networks within the cervical spinal cord can be transcutaneously neuromodulated to physiological states that enable and amplify voluntary control of the arm and hand

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over, both sexes.
* At least 6 weeks post-implant (in participants having a surgery for an implant to stabilise the spine).
* ISNCSCI upper extremity motor score between 5 and 30 (both arms/hands)
* GRASSP-strength score >=15 & <70
* Medically stable, cognitively intact and able to breathe independently.
* Attending upper limb therapy sessions at the QENSIU
* Planned stay longer than the duration of the intervention
* Able to sit for more than 2 hours a day

Exclusion Criteria:

* Unstable cervical spine injury
* Needing ventilation assistance during daytime
* Any implanted active metallic device without unconfirmed MRI compatibility (in our previous studies, we safely applied tESCS to participants with MRI-compatible devices/implants)
* Pregnancy and/or lactation.
* Non-injury-related neurological impairment
* Severe spasticity which have been unstable prior to enrolment
* Botulinum toxin injections-
* Clinically significant severe depression
* Patients who have cardiovascular disease
* Patients with severe ongoing Autonomic Dysreflexia
* Skin conditions or allergies that may affect electrode placement.
* Current infections
* Patients who have been involved in any other interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Retention | From enrollment till the last assesment at 8 weeks
  Recruitment and retention
Interference | From enrolment till the end of intervention at 4 weeks
  Interference with daily routine
Stimulation | From the first till the last intervention session at 4 weeks
  Optimal current stimulation intensity in mA
Adverse effects | from the first till the last intervention session at 4 weeks
  The number of adverse effects
Feedback | From enrolment till the last assesment at 8 weeks
  Semi structured interview

SECONDARY OUTCOMES:
Hand function | From the first intervention session till the last assesment at 8 weeks
  Sensory and motor test Graded and Redefined Assessment of Strength, Sensibility and Prehension (GRASSP), range 0-166 (0 no function, 116 all normal)
Spinal Cord Independence Measure | From the recruitment till the last assessment at 8 weeks
  Spinal Cord Independence Measure (range 0-100, 100 max independence)
Quality of life basic dataset | From recruitment till the last assessment at 8 weeks
  International Spinal Cord Injury Data Sets Quality of Life Basic Data Set -Data Form
Spasticity | From the enrolment till the last assesment at 8 weeks
  Modified Ashworth Scale range 0-4 (0 no increased tone, 4 very rigid)
Dynamometry | From the enrolment till the last assesment at 8 weeks
  Grip force
International Standard for Neurological Classification of Spinal Cord Injury | From the enrolment till the last assesment at 8 weeks
  International Standard for Neurological Classification of Spinal Cord Injury
Motor evoked potential | From the recruitment till the last assesment at 8 weeks
  Transcranial magnetic stimulation with EMG measurement of affected muscle response
Somato sensory evoked potential | From the recruitment till the last assesment at 8 weeks
  Measurement of the integrity of the sensory pathways
Muscle synergy | From the recruitment till the last assesments at 8 weeks
  Measurement of electromyography of muscles or the same arm/hand
Box and Block test (the number of transferred blocks in 60s, out of 150 blocks) | From the recruitment till the last assessment at 8 weeks
  Manual dexterity

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Vuckovic University O VUCKOVIC, PhD Biomed Eng, Study Director — School of Engineering, University of Glasgow; Mariel A Purcell, MB CHB BAO, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only for patients who agree to share the data. Electrophysiological data -motor evoked potential, somatosensory evoked potential
Supporting Information: Study Protocol, ICF
Time Frame: 1st January 2029
Access Criteria: Researchers contacting Professor Vuckovic or Dr Purcell. Data will not be publicly available on any site
URL: https://www.digihealthcare.scot/app/uploads/2023/08/Intra-NHS-Scotland-Information-Sharing-Accord-2023.pdf

REFERENCES:
- [Background] Han B, Enas NH, McEntegart D. Randomization by minimization for unbalanced treatment allocation. Stat Med. 2009 Nov 30;28(27):3329-46. doi: 10.1002/sim.3710. PMID 19739238
- [Background] Eldridge SM, Costelloe CE, Kahan BC, Lancaster GA, Kerry SM. How big should the pilot study for my cluster randomised trial be? Stat Methods Med Res. 2016 Jun;25(3):1039-56. doi: 10.1177/0962280215588242. Epub 2015 Jun 12. PMID 26071431
- [Background] Gawne F, Massey S, Duffell L. The Neurophysiological Effects of Cervical Transcutaneous Spinal Cord Stimulation With and Without a High Frequency Carrier in Able-Bodied Adults. Artif Organs. 2025 Jun 3. doi: 10.1111/aor.15031. Online ahead of print. PMID 40457929
- [Background] Salvador-De La Barrera S, Mora-Boga R, Ferreiro-Velasco ME, Seoane-Pillado T, Montoto-Marques A, Rodriguez-Sotillo A, Pertega Diaz S. A validity study of the Spanish-World Health Organization Quality of Life short version instrument in persons with traumatic spinal cord injury. Spinal Cord. 2018 Oct;56(10):971-979. doi: 10.1038/s41393-018-0139-2. Epub 2018 May 23. PMID 29795170
- [Background] Kirshblum SC, Burns SP, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Mulcahey MJ, Schmidt-Read M, Waring W. International standards for neurological classification of spinal cord injury (revised 2011). J Spinal Cord Med. 2011 Nov;34(6):535-46. doi: 10.1179/204577211X13207446293695. No abstract available. PMID 22330108
- [Background] McNicol EL, Osuagwu B, Purcell M, McCaughey EJ, Lincoln C, Cope L, Vuckovic A. Neurophysiological Effect of Transcutaneous Electrical Spinal Cord Stimulation in Chronic Complete Spinal Cord Injury. Artif Organs. 2025 Jun 30. doi: 10.1111/aor.15050. Online ahead of print. PMID 40583777
- [Background] Moritz C, Field-Fote EC, Tefertiller C, van Nes I, Trumbower R, Kalsi-Ryan S, Purcell M, Janssen TWJ, Krassioukov A, Morse LR, Zhao KD, Guest J, Marino RJ, Murray LM, Wecht JM, Rieger M, Pradarelli J, Turner A, D'Amico J, Squair JW, Courtine G. Non-invasive spinal cord electrical stimulation for arm and hand function in chronic tetraplegia: a safety and efficacy trial. Nat Med. 2024 May;30(5):1276-1283. doi: 10.1038/s41591-024-02940-9. Epub 2024 May 20. PMID 38769431
- [Background] Barss TS, Parhizi B, Porter J, Mushahwar VK. Neural Substrates of Transcutaneous Spinal Cord Stimulation: Neuromodulation across Multiple Segments of the Spinal Cord. J Clin Med. 2022 Jan 27;11(3):639. doi: 10.3390/jcm11030639. PMID 35160091
- [Background] Chandrasekaran S, Bhagat NA, Ramdeo R, Ebrahimi S, Sharma PD, Griffin DG, Stein A, Harkema SJ, Bouton CE. Targeted transcutaneous spinal cord stimulation promotes persistent recovery of upper limb strength and tactile sensation in spinal cord injury: a pilot study. Front Neurosci. 2023 Jul 7;17:1210328. doi: 10.3389/fnins.2023.1210328. eCollection 2023. PMID 37483349
- [Background] McGeady C, Vuckovic A, Singh Tharu N, Zheng YP, Alam M. Brain-Computer Interface Priming for Cervical Transcutaneous Spinal Cord Stimulation Therapy: An Exploratory Case Study. Front Rehabil Sci. 2022 Jun 23;3:896766. doi: 10.3389/fresc.2022.896766. eCollection 2022. PMID 36188944
- [Background] Inanici F, Samejima S, Gad P, Edgerton VR, Hofstetter CP, Moritz CT. Transcutaneous Electrical Spinal Stimulation Promotes Long-Term Recovery of Upper Extremity Function in Chronic Tetraplegia. IEEE Trans Neural Syst Rehabil Eng. 2018 Jun;26(6):1272-1278. doi: 10.1109/TNSRE.2018.2834339. PMID 29877852
- [Background] Freyvert Y, Yong NA, Morikawa E, Zdunowski S, Sarino ME, Gerasimenko Y, Edgerton VR, Lu DC. Engaging cervical spinal circuitry with non-invasive spinal stimulation and buspirone to restore hand function in chronic motor complete patients. Sci Rep. 2018 Oct 19;8(1):15546. doi: 10.1038/s41598-018-33123-5. PMID 30341390
- [Background] Gad P, Lee S, Terrafranca N, Zhong H, Turner A, Gerasimenko Y, Edgerton VR. Non-Invasive Activation of Cervical Spinal Networks after Severe Paralysis. J Neurotrauma. 2018 Sep 15;35(18):2145-2158. doi: 10.1089/neu.2017.5461. PMID 29649928
- [Background] Khorasanizadeh M, Yousefifard M, Eskian M, Lu Y, Chalangari M, Harrop JS, Jazayeri SB, Seyedpour S, Khodaei B, Hosseini M, Rahimi-Movaghar V. Neurological recovery following traumatic spinal cord injury: a systematic review and meta-analysis. J Neurosurg Spine. 2019 Feb 15;30(5):683-699. doi: 10.3171/2018.10.SPINE18802. Print 2019 May 1. PMID 30771786
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628